CLINICAL TRIAL: NCT01853189
Title: Effectiveness of Osteopathic Manipulative Treatment in Pediatric Asthma
Acronym: OMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OAsPed-1
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Asthma
Keywords: pediatrics; asthma; osteopathic manipulative treatment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMT + Usual Care (Other)
  Interventions: Other: OMT + Usual Care
- Usual Care (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: OMT + Usual Care — patients from this group received 6 sessions of OMT
  Arms: OMT + Usual Care
Other: Usual Care — patients from control group received standard care + osteopathic evaluation only, according to the same schedule of the study group
  Arms: Usual Care

SUMMARY:
Asthma is a highly prevalent chronic disease in children. Complementary and Alternative Medicine research on asthma showed a potential effect on pediatric patients.

Studies looking at the effect of Osteopathic Manipulative Treatment seems to reveal positive results.

The aim of study is to further explore the role of OMT on asthma in a pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* children with asthma age between 5 and 14

Exclusion Criteria:

* associated co-morbities surgical patients

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Difference in Forced expiratory volume in the 1st second (FEV1) before and after OMT | Participants will be assessed at entry, after 3 and 6 months.

SECONDARY OUTCOMES:
Difference in fractional exhaled nitric oxide (FeNO) before and after OMT | Participants will be assessed at entry, after 3 and 6 months.
Difference in percentage of hemoglobin saturation before and after OMT | Participants will be assessed at entry, after 3 and 6 months.
Difference in Pediatric Asthma Quality of Life Questionnaire (PAQOL) before and after OMT | Participants will be assessed at entry, after 3 and 6 months.
Differences in the number, type and quality of somatic dysfunctions | Participants will be assessed at entry, after 3 and 6 months
Difference in peak expiratory flow (PEF) before and after OMT | Participants will be assessed at entry, after 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Santo Spirito Hospital, Pescara, Abruzzo, Italy